CLINICAL TRIAL: NCT02454114
Title: HOME FIRST (HOME Followed - up With Infection Respiratory Support Team)
Brief Title: HOME FIRST Pilot: a Study of Early Supported Discharge in Patients With Lower Respiratory Tract Infections
Acronym: HOMEFIRST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12/NW/0731
Record Dates: First submitted 2015-05-08; First posted 2015-05-27 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2012-10

CONDITIONS: Community Acquired Pneumonia; Hospital Acquired Pneumonia; Lower Respiratory Tract Infection
Keywords: Pneumonia; Community; Hospital; Respiratory; Infection
MeSH Terms: conditions — Community-Acquired Pneumonia; Healthcare-Associated Pneumonia; Pneumonia; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Hospital Care (SHC) (Active Comparator): All management and discharge decisions will be made by the patient's usual hospital team. Clinical tests will be performed at the discretion of the medical team. If any significant or concerning clinical issues are noted during study team's visits, the usual medical team will be alerted. Patients receiving SHC will be discussed at weekly case note MDT meeting and followed-up on discharge in the 'Respiratory Infection' out-patient clinic (in the patient's own home if necessary) at 6 weeks, with a repeat chest X-ray if needed.
  Interventions: Other: Standard Hospital Care
- HOMEFIRST (Active Comparator): Patients randomised to HOMEFIRST care will initially receive up to twice daily visits for the first 48 hours. After this, the frequency and duration of visits will depend on clinical need but not exceed 5 days. The study nurse will establish the need for the involvement of other MDT members. Laboratory tests will be performed as clinically indicated. Venepuncture will be performed for clinical purposes as needed.
  Patients will be discussed at a weekly case-note MDT meeting and followed-up on discharge in the 'Respiratory Infection' out-patient clinic (in the patient's own home if necessary) at 6 weeks, with a repeat chest X-ray if needed.
  Patients are either discharged from HOMEFIRST, readmitted or handed over to their community care team at the end of the intervention.
  Interventions: Other: HOMEFIRST

INTERVENTIONS:
Other: HOMEFIRST — HOMEFIRST patients receive monitoring and review of; vital signs, symptoms, mental state, nutrition and hydration, urine output, skin turgor and integrity, mobility, coping ability, medication concordance, smoking and nutrition and hydration. Individualised verbal and written self-management plans, a list of symptoms (including red flag symptoms) to prompt contact with the study team and a 24hr emergency contact number are provided. Clinical bloods and other investigations will be taken/requested as necessary. Questionnaires will be completed as follows; SF-12 - at recruitment and 6 weeks, CAP-SYM - at recruitment and 6 weeks. Satisfaction questionnaires are conducted over the telephone at 2 wks by an independent assessor. As part of usual clinical practice patients will have bloods and radiology requested as required.
  Arms: HOMEFIRST
Other: Standard Hospital Care — No research investigations will occur except for questionnaires; as part of usual clinical practice patients will have bloods and radiology requested as desired by their usual clinical team.
  SF-12 (physical and mental function) [performed twice in total] - at recruitment (day 0) and 6 weeks
  CAP-SYM [performed 3 times in total] - at recruitment day 0 (twice including day minus 30) and 6 weeks
  Patient (and carer/consultee) satisfaction - conducted over the telephone at 2 wks by an independent assessor.
  Arms: Standard Hospital Care (SHC)

SUMMARY:
HOME FIRST (Home Followed - up with Infection Respiratory Support Team) is an early supported discharge scheme. It will enable patients with lower respiratory tract infection (LRTI) to be provided with high quality safe, effective, efficient patient centred care, tailored to their needs in their own home; aiming to improve the overall experience of the service user, improve patient outcomes and reduce hospital length of stay whilst simultaneously reducing admission rates, an area of major strategic importance to the NHS.

DETAILED DESCRIPTION:
A randomised interventional clinical care pathway study of early supported discharge (termed 'HOME FIRST') versus standard hospital care for patients hospitalised with LRTI.

HOME FIRST will provide co-ordinated multidisciplinary team (MDT) care, provision of 24hr emergency telephone cover, access to fully trained respiratory study nurse(s) and study doctor(s). The HOME FIRST MDT consists of:

* Study doctors (trained respiratory physicians - consultants and senior SpRs)
* Highly trained respiratory specialist nursing staff
* Close links with a physiotherapist (mobility and respiratory)
* Home help provision (temporary assistance with ADLs by carers) which may include occupational therapy or social worker involvement (HOME FIRST has fast access to meals-on-wheels)
* Close links with pharmacy for rapid dispensing of discharge medication.

Patients hospitalised with LRTI at the Royal Liverpool and Broadgreen (RLBUHT) Teaching Hospitals between October 2012 and April 2014 will be approached.

Patients (or the next of kin if the patient is unable to give informed consent) will be offered participation in the study if they fit the strict inclusion/exclusion criteria. They will be then be randomised to receive HOME FIRST or standard hospital care (SHC). The investigators will aim to recruit 25 patients to each arm of the study.

Patients randomised to HOME FIRST care will initially receive up to twice daily respiratory specialist nurse visits for the first 48 hours. After this time period, the frequency and duration of visits will depend on clinical need. The study nurse will establish the need for the involvement of other MDT team members. Laboratory tests will be performed as clinically indicated at the discretion of the study team. Venepuncture will be performed by fully trained research staff for clinical purposes as needed in the HOME FIRST limb: as for those patients in the SHC limb frequency of venepuncture depends on clinical assessment of need by their regular medical team.

Patients randomised to standard hospital care (SHC) - All management and discharge decisions will be made by the patient's usual hospital team. Clinical tests will be performed at the discretion of the medical team. If any significant or concerning clinical issues are noted during study team's visits, the usual medical team will be alerted.

All patients will be discussed at a weekly case-note MDT meeting. All patients will be followed-up on discharge in the 'Respiratory Infection' out-patient clinic (in the patient's own home if necessary) at 6 weeks, with a repeat chest X-ray if needed.

ELIGIBILITY:
Eligibility - Patients with any of the following conditions;

* Pneumonia - community-acquired (CAP) or hospital-acquired (HAP) - pneumonia definition - a series of clinical symptoms with radiological consolidation N.B. All pneumonia CURB-65 scores will be considered but patients with CURB-65 ≥3 MUST have had at least 24hrs of in-patient observation before recruitment into part B of the study.
* Pneumonia with concomitant COPD or bronchiectasis
* Non-pneumonic lower respiratory tract infection without COPD or bronchiectasis

Inclusion Criteria:

* Age>18yrs old
* All observations must be stable for 12-24hrs
* EWS ≤2 AND SBP>90 (all observations must be stable for 12-24hrs)
* Has a telephone
* Can manage activities of daily living with current available support (If needed, immediate occupational therapy/physiotherapy/social assessment and care can be arranged prior to discharge and continued at home)
* Improving/stable inflammatory markers
* Improving/stable U&Es
* Fluent English speaker

Exclusion Criteria;

* Acute exacerbations of COPD
* Acute exacerbations of bronchiectasis without consolidation
* Patients with CURB-65 >3 admitted <24 hours ago
* Patients unable to manage at home even with maximal support from HOME FIRST (This may include intravenous drug users, patients with history of excess alcohol consumption or mental health problems)
* Empyema or untapped pleural effusion (If no diagnostic pleural tap performed - discuss with study doctor)
* Serious co-morbidities requiring hospital treatment (e.g. CKD, CCF) or deemed unstable (significant AKD)
* Suspected MI/raised TnI/T consistent with NSTEMI (Or acute ECG changes) within 5 days of discharge
* Empyema or complicated parapneumonic effusion
* SBP<90mmHg
* Neutropenia
* No fixed abode
* Tuberculosis suspected
* Well enough for discharge without HOME FIRST support
* Oxygen saturations <92% on air - for patients without chronic respiratory illness Oxygen saturations <88% on air - for patients with chronic respiratory illness (excluding asthma for which oxygen saturations must be >92% on air). All such cases MUST be discussed as oxygen assessment may be needed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Time to recovery | Six weeks
  Our primary endpoint is time to recovery. This is assessed by our simple 'RECRTI' (functional RECovery from Respiratory Tract Infection) questionnaire (non-validated) which is completed at 6 weeks Patients (or consultees) will be asked at recruitment to define their/the patient's best exercise capacity in the last 3 months e.g chair to bed with 1, unlimited exercise tolerance etc
  At the 6 week out-patient appointment they will be asked 4 simple questions: (marked on a likert-type scale in days and weeks):
  1. When (if at all) did your sleep return to normal?
  2. When (if at all) did your diet/appetite return to normal?
  3. When (if at all) did your (pre-defined) exercise capacity return to normal?
  4. When (if at all) did your capacity to work or socialise (delete as appropriate) return to normal?
  With regards to the primary outcome of time to recovery, this is a non-inferiority trial.

SECONDARY OUTCOMES:
30-day mortality | up to 6 weeks after recruitment
  We will assess safety i.e. ensure there is no increase in mortality in the HOME FIRST limb.
30-day hospital readmission rates | up to 6 weeks after recruitment
  We will assess safety i.e. ensure there is no delayed recovery, no pneumonia (or non-pneumonia) complications resulting in hospital admission in the HOME FIRST arm.
Patient satisfaction using a validated satisfaction questionnaire | at 2 weeks post recruitment
  A validated patient satisfaction will be conducted at 2 weeks by an independent assessor.
Carer (NOK) satisfaction using a validated satisfaction questionnaire | at 2 weeks post recruitment
  A validated carer/consultee satisfaction will be conducted at 2 weeks by an independent assessor.
Length of stay in hospital | Participants will be followed for the duration of hospital stay, this may be 1 day to 1 year
  Length of hospital stay will be calculated.
Functional status as assessed by SF-12 validated questionnaire | up to 6 weeks after recruitment
  Functional status (physical and mental) and quality of life (QOL) questionnaire will be completed to assess recovery / post respiratory infection.
Pneumonia score as assessed by CAP-SYM validated questionnaire | up to 6 weeks after recruitment
  The questionnaire will be completed to assess recovery / post respiratory infection
Combined total length of stay (days) - hospital and home first | Participants will be followed for the duration of hospital stay and their HOME FIRST stay, the latter can range from 1 - 5 days
  Total length of stay - combined will be calculated

OTHER OUTCOMES:
Health - economic | One year
  A formal planned health economic analysis (by an NIHR Research Design Service [RDS] recommended health-economist) will measure costs and resource utilisation, using costs that are sensitive to the different resources used during each care episode, to assess the cost-effectiveness of HOME FIRST.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen B Gordon, Professor, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Royal Liverpool And Broadgreen University Hospital, Liverpool, Merseyside, United Kingdom